CLINICAL TRIAL: NCT01027455
Title: Warm Humidified Insufflation for Laparoscopic Appendicectomy in Children: a Randomised Controlled Trial
Brief Title: Warm Humid Gas Insufflation for Appendix Removal by Minimally Invasive Surgery Warm Humid Insufflation for Appendix Removal by Minimally Invasive Surgery Trial (WARMIST)
Acronym: WARMIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Auckland District Health Board (Other Government)
Responsible Party: Mr James KM Hamill, Auckland District Health Board
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WARMIST
Record Dates: First submitted 2009-12-07; First posted 2009-12-08 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2009-10

CONDITIONS: Peritoneal Dessication Damage and Inflammation; Peri-operative Hypothermia
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dry Cold (Placebo Comparator): Dry (0% relative humidity) and cold (20 degrees Celsius - Room Temperature) carbon dioxide gas intraperitoneal insufflation for laparoscopic appendicectomy
  Interventions: Procedure: Laparoscopic Appendicectomy
- Humidification (Experimental): Humidified (98% relative humidity) and warm (37 degrees Celsius) carbon dioxide gas intraperitoneal insufflation for laparoscopic appendicectomy
  Interventions: Device: Fisher and Paykel Insuflow (MR 860) Surgical Humidification Device; Procedure: Laparoscopic Appendicectomy

INTERVENTIONS:
Device: Fisher and Paykel Insuflow (MR 860) Surgical Humidification Device — Humidified warm carbon dioxide gas insufflation during laparosopic procedure
  Arms: Humidification
Procedure: Laparoscopic Appendicectomy — Dry and Cold carbon dioxide gas insufflation
  Arms: Dry Cold
Procedure: Laparoscopic Appendicectomy — Humidified warm carbon dioxide gas insufflation during laparosopic procedure
  Arms: Humidification

SUMMARY:
In laparoscopic (key-hole) surgery, the use of cold dry carbon dioxide gas to inflate the abdominal cavity for the creation a clear operating field, results in damage to the cavity lining, known as the peritoneum. This has been associated with negative effects on post-operative recovery. Adult studies using warm humidified insufflation gas have indicated possible decreased post-operative pain, reduced narcotic analgesia requirements, decreased fogging of the laparoscopic camera lens, and reduced time to return to normal activities. Cold dry gas during laparoscopic surgery also has potential to cause abnormal decrease in body core temperature (hypothermia). This has been established by trials in adult humans and animal models. The WARMIST study aims to investigate for whether warm humid gas insuflation during laparoscopic removal of the appendix in children reduces intraoperative temperature variations, post-operative pain (indicated by morphine usage and pain scores), length of hospital stay and degree of camera lens fogging, and speed post-operative recovery compared to using cold dry gas insufflation.

DETAILED DESCRIPTION:
Study Aim/Question:

Does warm humidified carbon dioxide gas compared to cold dry gas for abdominal cavity insufflation during laparoscopic appendectomy in children reduce variations in intraoperative core body temperature, reduce post-operative pain, and improve post-operative recovery?

The Aim of this study is to investigate whether differences exist in the following outcomes:

1. Intraoperative temperature variation;
2. Need for post-operative opiate analgesia (primary outcome of the study);
3. Post-operative pain scores;
4. Length of hospital stay;
5. Post-operative return to normal daily activities;
6. Fogging of laparoscope lens; when warm humidified rather than cold dry gas is used for intra-abdominal insufflation during laparoscopic appendectomy for acute appendicitis in children.

Study Sample Size and Power Calculations:

From a retrospective audit of 43 children who underwent laparoscopic appendicectomy at Starship Children's Hospital in 2006, 70% required opiate-based analgesia for pain relief during some stage of their admission. To detect a 30% reduction from 70% (i.e. 49% of the exposure group will require opiates) with power of 0.8 and alpha of 0.05 using 2 tailed Fisher's exact test, 95 participants will be needed per arm of the trial.

Study Participants:

* Inclusion criteria:

Children aged 8-14 years presenting to Starship Children's Hospital within the study period diagnosed clinically with acute appendicitis requiring diagnostic laparoscopy +/- appendicectomy.

* Exclusion criteria:

Consent to participate in study not obtained, partial or total blindness, unable to speak and read sufficient English, presence of any abdominal prostheses, diagnosis of mental retardation, developmental delay, neuro-muscular impairment, attention-deficit disorder, chronic pain, or psychiatric illness, immunosuppression, allergy to morphine, and history of previous abdominal surgery.

Study Design:

This is a Randomised-Controlled Trial involving 190 children aged between 8-14 years presenting to Starship Children's Hospital with clinical signs of acute appendicitis. After recruitment, study participants will be randomised to either the intervention group (warm humidified gas insufflation) or control group (cool dry gas insufflation) before undergoing laparoscopic appendicectomy as part of the surgical management of acute appendicitis. The insufflation device used will the the Fisher and Paykel Insuflow MR 860. Other intraoperative variables will be controlled or standardised.

A computer-generated random sequence will be employed to randomise study participants. Group allocations will be placed in sealed opaque envelopes and these will be opened in sequence for consecutive participants. Allocations will be concealed until completion of data collection. To ensure double-blinding (blinding of investigators, operating surgeons, members of the clinical team, study participants and family), circulating theatre nurses who have no direct involvement in the care of participants will be unblinded and control the switches to the insufflation device. Upon opening an allocation envelope, they will set the Insuflow device on warm humidified or cold dry gas insufflation and place a specially designed cover over the device before transferring the device into the operating theatre. This cover will be placed over the insufflation device for the duration of the operation to blind other theatre personnel. At the end of the operation, the insufflation device will be switched off and removed from theatre by circulating theatre nurses with the cover intact. It will be disassembled in the theatre preparation room, out of sight.

The following data will be measured/collected intraoperatively:

1. Core body temperature measured every 10 minutes from a nasogastric temperature probe, placed after anaesthetic induction;
2. Severity of laparoscopic camera lens fogging: Surgeon's rating of the severity of camera fogging (scale of 1 to 10 - 10 representing worst degree of fogging);
3. Surgeon's rating of the operation's technical difficulty (scale of 1 to 10 - 10 representing most difficult);
4. Total volume of CO2 gas used for pneumoperitoneum creation and maintenance;
5. Duration of operation;
6. Total amount of analgesia and anti-emetics given intraoperatively;
7. Pathological appearance of appendix and degree of peritoneal faecal/pus contamination if appendix perforation is present;
8. Temperature and volume of intravenous fluids administered and any peritoneal irrigation fluids used.

A standard perioperative care protocol will be used to ensure all study patients receive the same standard of care, reducing risk of performance bias. The protocol will cover perioperative use of antibiotics, measures to prevent infections including wound infections, post-operative oral feeding and mobilisation, criteria for discharge, etc.

Post-operative opioid-sparing analgesia medication (paracetamol and non-steroidal anti-inflammatory agents) will be standardised for all study participants in the post-anaesthesia care unit (PACU) and on the surgical ward. The route of administration will depend on the degree of nausea and vomiting, with both oral and per rectal preparations available.

A Visual Analogue Scale (VAS) from 0 to 10 will be used to measure pain and to ascertain requirements for additional nurse-controlled analgesia. All opiate-based analgesia required in the first 12 hours post-operatively will be administered intravenously to minimize variations in gastrointestinal absorption and effects of post-operative nausea and vomiting (PONV).

The following outcomes will be measured and recorded post-operatively:

1. Tympanic body temperature at 10-minute intervals for the duration of stay in PACU
2. Presence of shivering in PACU
3. Post-operative pain scores at rest and with movement, measured using 10-point pictorial Visual Analogue Scale (VAS)at the following times: 2, 4, 6, 8, 10, 12, 24, and 48 hours from end of operation.
4. Total Nurse-controlled Opioid Analgesia required, both oral and parenteral, converted to Mean Equivalent Daily Dose (MEDD) units of parenteral morphine, in the first 12, 24 and 48 hours post-operatively and during the entire hospital stay.

   The need for opioid analgesia and the total quantity required for the total duration of hospital stay will be the primary outcome for this study.

   The opiate-based analgesia available for this study are: oral morphine, IV morphine, and IV fentanyl.
5. Severity of post-operative nausea, number of vomiting episodes and total amount of anti-emetic medications required.
6. Total length of laparoscopic port site wounds, measured in millimetres during the first dressing change
7. Length of hospital stay (days)
8. Post-operative return of normal activities is measured using a Day-10 Post-operative Recovery Questionnaire given to participants and family at the time of discharge from hospital. Participants are asked to complete this questionnaire the morning of Day 10 after their operation and post it back to the investigators in a pre-paid envelope provided. The Questionnaire is adapted from the Pediatric Quality of Life Inventory Version 4.0. The Principle Investigator will remind participants with a phone call one to two days before the Questionnaire has to be completed.

All operative and disease-related complications (minor and major) during hospital stay or reported at the follow-up outpatient clinic will also be recorded. Standard internationally-recognized definitions of operative complications will be used.

Statistical Analysis of Data:

Intervention and Control groups will be compared using Fisher's exact test for categorical variables and appropriate non-paired parametric or non-parametric statistical tests for continuous variables, depending of the normality of the data. Statistical significance will be set at 2-tailed P value <.05.

Subgroup analysis of the uncomplicated and complicated appendicitis groups will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 8-14 years presenting to Starship Children's Hospital (Auckland, New Zealand) within the study period diagnosed clinically with acute appendicitis requiring diagnostic laparoscopy +/- appendicectomy.

Exclusion Criteria:

* Consent to participate in study not obtained, partial or total blindness, unable to speak and read sufficient English, presence of any abdominal prostheses, diagnosis of mental retardation, developmental delay, neuromuscular impairment, attention-deficit disorder, chronic pain, or psychiatric illness, immunosuppression, allergy to morphine, and history of previous abdominal surgery

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 190 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Post-operative Morphine equivalent analgesia use | PACU, Post-operative 12 hours, Post-operative 24 hours, Post-operative 48 hours, Duration of hospital stay
Peri-operative Core Body Temperature Variation | Intra-operative, Duration of stay in PACU

SECONDARY OUTCOMES:
Pain scores measured by Visual Analogue Scale | Pre-operative baseline and Post-operative 2, 4, 6, 8, 10, 12, 24, 48 hours
Post-operative Return to Normal Daily Activities | Post-operative Day 10 Recovery Questionnaire
Severity of Post-operative Nausea and Vomiting as indicated by Antiemetic use | Post-operative Day 0, Day 1, Day 2, Day 3
Peri-operative Complications (operative and disease-related) | Up to 6 weeks post-operatively
Severity of Laparoscopic Camera Lens Fogging | Intra-operative

CONTACTS AND LOCATIONS:
Locations (1):
- Starship Children's Hospital, Auckland, New Zealand

REFERENCES:
- [Derived] Yu TC, Hamill JK, Liley A, Hill AG. Warm, humidified carbon dioxide gas insufflation for laparoscopic appendicectomy in children: a double-blinded randomized controlled trial. Ann Surg. 2013 Jan;257(1):44-53. doi: 10.1097/SLA.0b013e31825f0721. PMID 22824858